CLINICAL TRIAL: NCT04742738
Title: A 2-Stage, Phase I/II, Placebo-controlled, Randomized, Observer-blinded, Dose-finding Study to Assess the Safety, Reactogenicity, and Immunogenicity of a SARS-CoV-2 Recombinant Protein Nanoparticle Vaccine (GBP510) Adjuvanted With Aluminum Hydroxide in Healthy Younger and Older Adults
Brief Title: Safety and Immunogenicity Study of SARS-CoV-2 Nanoparticle Vaccine (GBP510) Adjuvanted With Aluminum Hydroxide (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SK Bioscience Co., Ltd. (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GBP510_001
Record Dates: First submitted 2021-02-04; First posted 2021-02-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 (Healthy Volunteers)
MeSH Terms: conditions — COVID-19 | interventions — aluminum sulfate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Test group 1 - Stage 1 Low dose-level Cohort (Experimental): 2 doses of GBP510 adjuvanted with Alum (Receptor Binding Domain (RBD) 10μg/dose), 1 dose each on Days 0 and 28.
  Interventions: Biological: GBP510 adjuvanted with Alum (RBD 10μg/dose) - Stage 1
- Placebo group - Stage 1 Low dose-level Cohort (Placebo Comparator): 2 doses of Placebo Saline, 1 dose each on Days 0 and 28.
  Interventions: Other: Normal saline (0.9% sodium chloride solution) - Stage 1
- Test group 2 - Stage 1 High dose-level Cohort (Experimental): 2 doses of GBP510 adjuvanted with Alum (RBD 25μg/dose), 1 dose each on Days 0 and 28.
  Interventions: Biological: GBP510 adjuvanted with Alum (RBD 25μg/dose) - Stage 1
- Placebo group - Stage 1 High dose-level Cohort (Placebo Comparator): 2 doses of Placebo Saline, 1 dose each on Days 0 and 28.
  Interventions: Other: Normal saline (0.9% sodium chloride solution) - Stage 1
- Test group 1 - Stage 2 (Experimental): 2 doses of GBP510 adjuvanted with Alum (RBD 10μg/dose), 1 dose each on Days 0 and 28.
  Interventions: Biological: GBP510 adjuvanted with Alum (RBD 10μg/dose) - Stage 2
- Test group 2 - Stage 2 (Experimental): 2 doses of GBP510 adjuvanted with Alum (RBD 25μg/dose), 1 dose each on Days 0 and 28.
  Interventions: Biological: GBP510 adjuvanted with Alum (RBD 25μg/dose)- Stage 2
- Placebo group - Stage 2 (Placebo Comparator): 2 doses of Placebo Saline, 1 dose each on Days 0 and 28.
  Interventions: Other: Normal saline (0.9% sodium chloride solution)- Stage 2

INTERVENTIONS:
Biological: GBP510 adjuvanted with Alum (RBD 10μg/dose) - Stage 1 — Participants will receive intramuscular (IM) injections of GBP510 adjuvanted with Alum (RBD 10μg/dose) on Days 0 and 28.
  Other Names: GBP510-Alum-10μg
  Arms: Test group 1 - Stage 1 Low dose-level Cohort
Other: Normal saline (0.9% sodium chloride solution) - Stage 1 — Participants will receive intramuscular (IM) injections of Normal saline on Days 0 and 28.
  Arms: Placebo group - Stage 1 Low dose-level Cohort
Biological: GBP510 adjuvanted with Alum (RBD 25μg/dose) - Stage 1 — Participants will receive intramuscular (IM) injections of GBP510 adjuvanted with Alum (RBD 25μg/dose) on Days 0 and 28.
  Other Names: GBP510-Alum-25μg
  Arms: Test group 2 - Stage 1 High dose-level Cohort
Other: Normal saline (0.9% sodium chloride solution) - Stage 1 — Participants will receive intramuscular (IM) injections of Normal saline on Days 0 and 28.
  Arms: Placebo group - Stage 1 High dose-level Cohort
Biological: GBP510 adjuvanted with Alum (RBD 10μg/dose) - Stage 2 — Participants will receive intramuscular (IM) injections of GBP510 adjuvanted with Alum (RBD 10μg/dose) on Days 0 and 28.
  Other Names: GBP510-Alum-10μg
  Arms: Test group 1 - Stage 2
Biological: GBP510 adjuvanted with Alum (RBD 25μg/dose)- Stage 2 — Participants will receive intramuscular (IM) injections of GBP510 adjuvanted with Alum (RBD 25μg/dose) on Days 0 and 28.
  Other Names: GBP510-Alum-25μg
  Arms: Test group 2 - Stage 2
Other: Normal saline (0.9% sodium chloride solution)- Stage 2 — Participants will receive intramuscular (IM) injections of Normal saline on Days 0 and 28.
  Arms: Placebo group - Stage 2

SUMMARY:
This is a first-in-human, Phase I/II, randomized, placebo-controlled, observer-blinded, age-escalating study to assess the safety, reactogenicity and immunogenicity of a SK SARS-CoV-2 recombinant protein nanoparticle vaccine (GBP510) adjuvanted with Alum in healthy younger and older adults.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety, reactogenicity and immunogenicity of the candidate vaccine administered twice with 28-day interval in healthy adults including older adults.

A total of 260 healthy younger and older adults will be enrolled to receive 2 doses of either one GBP510 formulation (Test group 1 or 2) or placebo saline (Placebo group).

This study will consist of 2 stages, and a stepwise approach will be adopted as a safety precaution. Approximately 60 healthy adults aged 19 to 55 years will be enrolled and vaccinated first in Stage 1, and blinded safety data collected through 7 days after the last study vaccination will be reviewed by the sponsor, and then by the independent Data Safety Monitoring Board (DSMB) in an unblinded manner. Advancement to Stage 2 for further enrollment of 200 healthy younger and older adults aged 19 to 85 years will be determined if an acceptable safety profile is confirmed based on the sponsor and DSMB review. DSMB will recommend whether to proceed to the next stage or not, and DSMB may suggest discontinuation of the study or adjustment of dose and dosing regimen based on the safety review.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

Age

1. For Stage 1, participant must be 19 to 55 years of age inclusive, at the time of signing the informed consent.

   For Stage 2, participant must be 19 to 85 years of age inclusive, at the time of signing the informed consent

   Type of Participant and Disease Characteristics
2. Participants who are healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, and medical judgement of the investigator
3. Participants who are able to attend all scheduled visits and comply with all study procedures.

   Weight
4. Body mass index (BMI) within the range 18-30 kg/m2 at screening (inclusive)

   Sex and Contraceptive/Barrier Requirements
5. Female participants of childbearing potential must agree to be heterosexually inactive, or agree to consistently use at least one acceptable method of contraception from at least 4 weeks prior to the 1st study vaccination to 12 weeks after the last study vaccination
6. Female participants with a negative urine or serum pregnancy test at screening

   Informed Consent
7. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Any clinically significant respiratory symptoms (e.g. cough, sore throat), febrile illness (tympanic temperature >38°C), or acute illness within 72 hours prior to the 1st study vaccination. A prospective participant should not be included until 72 hours after the condition has resolved.
2. History of virologically-confirmed COVID-19 disease, or definite or suspected exposure to anyone known to have SARS-CoV-2 infection
3. History of virologically-confirmed SARS or MERS disease
4. History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease
5. Any positive test results for hepatitis B, C, or HIV at screening
6. History of bleeding disorder or thrombocytopenia which is contraindicating intramuscular vaccination in the investigator's opinion
7. History of hypersensitivity and severe allergic reaction (e.g. anaphylaxis, Guillain-Barre syndrome) to any vaccines or components of the study intervention
8. History of malignancy within 5 years prior to the 1st study vaccination
9. Significant chronic illness that, in the opinion of the investigator, might increase risk of severe COVID-19, or interfere with the evaluation of the study objectives (e.g. asthma, chronic pulmonary disease, cardiovascular disease, chronic liver disease, diabetes mellitus, uncontrolled hypertension, renal disorders)
10. History of, or planned surgery under general anesthesia from 1 year prior to the 1st study vaccination through the study period
11. Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g. neurologic or psychiatric conditions)
12. Female participants who are pregnant or breastfeeding
13. (Only for Stage 1) Current smokers or a recent smoking history within 12 weeks prior to the 1st study vaccination. Occasional smokers who smoke up to 10 cigarettes per month may be allowed to participate at the investigator's discretion

    Prior/Concomitant therapy
14. Receipt of any medications or vaccinations intended to prevent COVID-19.
15. Receipt of any vaccine within 4 weeks prior to the 1st study vaccination or planned receipt of any vaccine from enrollment through 28 days after the last study vaccination (Visit 7), except for influenza vaccination, which may be received at least 2 weeks prior to the 1st study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines
16. Receipt of immunoglobulins and/or any blood or blood products within 12 weeks prior to the 1st study vaccination
17. Chronic use (more than 2 consecutive weeks) of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) within 12 weeks prior to the 1st vaccination. The use of topical and nasal glucocorticoids will be permitted.

    Prior/Concurrent Clinical Study Experience
18. Participation in another clinical study involving study intervention within 6 months prior to the 1st study vaccination, or concurrent, planned participation in another clinical study with study intervention during this study period.

    Other Exclusions
19. Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.
20. Healthcare worker or emergency response personnel in an occupation with a high risk of exposure to SARS-CoV-2

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of immediate systemic reactions - Stage 1 | Through 30 minutes (2 hours for sentinel participants) post-vaccination
Occurrence of solicited local Adverse Events (AEs) during 7 days post each vaccination - Stage 1 | Through 7 days post-vaccination
Occurrence of solicited systemic AEs during 7 days post each vaccination - Stage 1 | Through 7 days post-vaccination
Occurrence of unsolicited AEs during 28 days post each vaccination - Stage 1 | Through 28 days post-vaccination
Occurrence of Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs) and Adverse Events of Special Interest (AESIs) during the whole study period - Stage 1 | Through Day 0 to Day 365 post last vaccination
(Only in Sentinel group) Occurrence of out-of-normal range clinical laboratory test results (including change from baseline values) during 7 days post 1st vaccination - Stage 1 | Through 7 days post 1st vaccination
GMT of IgG antibody to the SARS-CoV-2 RBD measured by Enzyme-linked Immunosorbent Assay (ELISA) - Stage 2 | Through Day 365 post last vaccination
GMFR of IgG antibody to the SARS-CoV-2 RBD from baseline measured by ELISA - Stage 2 | Through Day 365 post last vaccination
Percentage of participants with ≥ 4-fold rise from baseline in ELISA IgG titer - Stage 2 | Through Day 365 post last vaccination
GMT of neutralizing antibody to the SARS-CoV-2 measured by pseudovirus and wild-type virus neutralization assays - Stage 2 | Through Day 365 post last vaccination
GMFR of neutralizing antibody to the SARS-CoV-2 from baseline measured by pseudovirus and wild-type virus neutralization assays - Stage 2 | Through Day 365 post last vaccination
Percentage of participants with ≥ 4-fold rise from baseline in pseudovirus and wild-type neutralizing antibody titer - Stage 2 | Through Day 365 post last vaccination
Cell-mediated response for both Th1 and Th2 (e.g. INF-γ, IL-4 using Enzyme-linked ImmunoSpot (ELISpot) or other system) - Stage 2 | Through Day 28 post last vaccination

SECONDARY OUTCOMES:
GMT of IgG antibody to the SARS-CoV-2 RBD measured by ELISA - Stage 1 | Through Day 365 post last vaccination
GMFR of IgG antibody to the SARS-CoV-2 RBD from baseline measured by ELISA - Stage 1 | Through Day 365 post last vaccination
Percentage of participants with ≥ 4-fold rise from baseline in ELISA IgG titer - Stage 1 | Through Day 365 post last vaccination
GMT of neutralizing antibody to the SARS-CoV-2 measured by pseudovirus and wild-type virus neutralization assays - Stage 1 | Through Day 365 post last vaccination
GMFR of neutralizing antibody to the SARS-CoV-2 from baseline measured by pseudovirus and wild-type virus neutralization assays - Stage 1 | Through Day 365 post last vaccination
Percentage of participants with ≥ 4-fold rise from baseline in pseudovirus and wild-type neutralizing antibody titer - Stage 1 | Through Day 365 post last vaccination
Cell-mediated response for both Th1 and Th2 (e.g. INF-γ, IL-4 using ELISpot or other system) - Stage 1 | Through Day 28 post last vaccination
Occurrence of immediate systemic reactions - Stage 2 | Through 30 minutes (2 hours for elderly participants aged 75 years and older) post-vaccination
Occurrence of solicited local AEs during 7 days post each vaccination - Stage 2 | Through 7 days post-vaccination
Occurrence of solicited systemic AEs during 7 days post each vaccination - Stage 2 | Through 7 days post-vaccination
Occurrence of unsolicited AEs during 28 days post each vaccination - Stage 2 | Through 28 days post-vaccination
Occurrence of SAEs, MAAEs and AESIs during the whole study period - Stage 2 | Through Day 0 to Day 365 post last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Cheong, Principal Investigator — Korea University Guro Hospital
Locations (12):
- South Korea (12):
  - Korea University Ansan Hospital, Ansan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Ewha Womans University Medical Center, Seoul
  - Hallym University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ajou University Hospital, Suwon

REFERENCES:
- [Derived] Arunachalam PS, Walls AC, Golden N, Atyeo C, Fischinger S, Li C, Aye P, Navarro MJ, Lai L, Edara VV, Roltgen K, Rogers K, Shirreff L, Ferrell DE, Wrenn S, Pettie D, Kraft JC, Miranda MC, Kepl E, Sydeman C, Brunette N, Murphy M, Fiala B, Carter L, White AG, Trisal M, Hsieh CL, Russell-Lodrigue K, Monjure C, Dufour J, Spencer S, Doyle-Meyers L, Bohm RP, Maness NJ, Roy C, Plante JA, Plante KS, Zhu A, Gorman MJ, Shin S, Shen X, Fontenot J, Gupta S, O'Hagan DT, Van Der Most R, Rappuoli R, Coffman RL, Novack D, McLellan JS, Subramaniam S, Montefiori D, Boyd SD, Flynn JL, Alter G, Villinger F, Kleanthous H, Rappaport J, Suthar MS, King NP, Veesler D, Pulendran B. Adjuvanting a subunit COVID-19 vaccine to induce protective immunity. Nature. 2021 Jun;594(7862):253-258. doi: 10.1038/s41586-021-03530-2. Epub 2021 Apr 19. PMID 33873199